CLINICAL TRIAL: NCT00583817
Title: Endovascular Treatment of Thoracic Aortic Disease
Acronym: EVOLVE Aorta
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Matthew Eagleton (Other)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Sponsor-Investigator, Matthew Eagleton, Physician Sponsor/PI, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G000101; 2018P001301 (Other: Massachusetts General Hospital IRB); 2018P001300 (Other: Massachusetts General Hospital IRB); 2018P001299 (Other: Massachusetts General Hospital IRB)
Record Dates: First submitted 2007-12-20; First posted 2007-12-31 (Estimated); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Thoracic Aortic Aneurysms; Dissecting, Aneurysm; Ascending Aorta Aneurysm; Aortic Arch; Aneurysm, Dissecting; Ascending Aortic Dissection; Thoracoabdominal Aortic Aneurysm; Renal Artery Aneurysm; Superior Mesenteric Artery Aneurysm; Aortic Dissection
MeSH Terms: conditions — Aortic Aneurysm, Thoracic; Aortic Dissection; Aneurysm, Ascending Aorta; Aneurysm; Dissection, Ascending Aorta; Aortic Aneurysm, Thoracoabdominal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (3):
- Ascending Aortic Arm (Experimental): Investigational endovascular stent-graft implantation to exclude aneurysm or repair dissection of the ascending aorta.
  Interventions: Device: Endovascular stent-graft implantation
- Arch Branch Arm (Experimental): Investigational endovascular stent-graft implantation to exclude aneurysm or repair dissection of the aortic arch.
  Interventions: Device: Endovascular stent-graft implantation
- Thoracoabdominal Aortic Arm (Experimental): Investigational endovascular stent-graft implantation to exclude thoracoabdominal aortic pathology including aortic aneurysms, renal artery aneurysms, and superior mesenteric artery aneurysms.
  Interventions: Device: Endovascular stent-graft implantation

INTERVENTIONS:
Device: Endovascular stent-graft implantation — Endovascular repair of aorta
  Other Names: Arch Branched Device (Cook Medical); Custom Made Fenestrated/Branched Endovascular Device (Cook Medica); Helical Hypogastric Branched Device (Cook Medical); Ascending Aortic Endograft (Cook Medical)

SUMMARY:
The purpose of this study is to assess the role endovascular therapy to treat aortic disease involving the ascending aorta, the aortic arch, and the visceral segment of the aorta (or thoracoabdominal aorta)

DETAILED DESCRIPTION:
This study is a prospective, non-randomized, single-site evaluation of the use of novel endovascular technology to treat complex aortic disease.

In an effort to allow for the evaluation of patients with both complex anatomic condition and challenging physiologic situations there are three study subsections as follows:

1. Ascending Arm Protocol: The intended use of the study is to provide endovascular therapy to patients with ascending aortic pathology including aneurysm, pseudoaneurysm, and/or aortic dissection who are considered high risk for conventional surgery. This will involve disease in the aorta from the sinotubular junction to the innominate artery.
2. Aortic Arch Arm Protocol: The intended use of the study is to provide endovascular therapy to patients with aortic arch pathology including aneurysm, pseudoaneurysm and/or aortic dissection who are considered high risk for conventional surgery. This will involve disease in aorta from the sinotubular junction to descending thoracic aorta.
3. Thoracobabdominal Aortic Arm Protocol: The intended use of the study is to provide endovascular therapy to patients with thoracoabdominal aortic pathology including aortic aneurysms, renal aneurysms, and superior mesenteric artery aneurysms. This will involve the aorta from the left carotid artery origin through the iliac artery bifurcation.

In addition, the purpose of the study is also characterized based on the protocol arm that patients are enrolled:

1. Ascending Arm Protocol: The purpose of this study is to assess the safety, efficacy, and intermediate (or long-term) rupture free survival rate of high risk surgical patients undergoing endovascular repair of ASCENDING AORTIC pathology including aortic dissection, aortic aneurysm, and/or aortic pseudoaneurysm. The objectives of this arm are as follows:

   * To assess the safety, efficacy and intermediate (or long-term) durability of an endovascular prosthesis as a means of preventing ascending aortic growth and rupture in high risk patients.
   * To measure the physiologic effects and outcomes of endovascular aneurysm repair.
   * Establish selection criteria, improve device design, operative technique and follow-up procedures for patients undergoing endovascular aneurysm repair.
2. Arch Arm Protocol: The purpose of this study is to assess the safety, efficacy, and intermediate (or long-term) rupture free survival rate of high risk surgical patients undergoing endovascular repair of AORTIC ARCH pathology including aortic aneurysm, pseudoaneurysm and/or dissection. The objectives of this arm are as follows:

   * To assess the safety, efficacy and intermediate (or long-term) durability of an endovascular prosthesis as a means of preventing aortic arch growth and rupture in high risk patients.
   * To measure the physiologic effects and outcomes of endovascular aneurysm repair.
   * Establish selection criteria, improve device design, operative technique and follow-up procedures for patients undergoing endovascular aneurysm repair.
3. Thoracoabdominal Arm Protocol: The purpose of this study is to assess the long-term safety, durability and rupture free survival of surgical patients undergoing endovascular repair of the THORACOABDOMINAL AORTA involving pathologies that include thoracoabdominal aortic aneurysms, renal artery aneurysms and superior mesenteric artery aneurysms.

   * To assess the long-term safety and durability of an endovascular prosthesis as a means of preventing aneurysm growth and rupture in patients having aneurysms involving the THORACOABDOMINAL AORTA.
   * To measure the physiologic effects and outcomes of endovascular aneurysm repair.
   * Establish selection criteria, improve device design, operative technique and follow-up procedures for patients undergoing endovascular aneurysm repair involving the THORACOABDOMINAL AORTA.

ELIGIBILITY:
Ascending Arm Protocol:

1. General Inclusion Criteria (Must meet ALL of the following):

   * Life expectancy greater than 2 years
   * Suitable arterial anatomy
   * Absence of systemic disease or allergy that precludes an endovascular repair
   * Capable of giving informed consent and willingness to comply with follow up schedule
   * Patient is considered high or prohibitive risk for open surgical repair of the ascending aneurysm or dissection
2. Anatomic Inclusion Criteria

   * Have ONE of the following

     1. Focal aneurysm in ascending aorta
     2. Pseudoaneurysms and/or dissections that are distal to the sinotubular junction.
     3. A thoracoabdominal aortic aneurysm ≥ 5.0 cm in women and ≥ 5.5 cm in men
     4. Have morphology or growth suggestive of immanent rupture
   * Must meet ALL of the following:

     1. Proximal Fixation:

        1. >15 mm aortic length distal to a patent coronary artery or coronary artery bypass that are considered patent and necessary for proper cardiac perfusion.

           * Proximal fixation may occur in either native aorta or surgical graft
           * In the setting of the aortic dissection, the proximal fixation must be proximal to the entry tear.
           * In the setting of aortic dissection, true lumen size must be large enough to allow deployment of the device
        2. Aortic diameter at the sinotubular junction >20 mm and ≤ 38mm
     2. Distal Fixation: a length of distal ascending aorta >5mm proximal to the innominate artery whereby seal and fixation can be achieved (the dissection flap may transcend the arch, but the seal must be achievable within the true lumen of the dissection)

        1. Aortic diameter (true lumen diameter in the setting of a dissection) at the innominate artery is ≤ 42mm. If the diameter at the innominate artery is ≥ 38mm the Low Profile version must be used
        2. Distance from the ascending aorta to the innominate artery must be >35mm
   * Iliac artery access

     1. Iliac anatomy must allow for the delivery of the endograft device which is loaded within an 18F-24F sheath.
     2. Conduits to the iliac vessels or aorta may be used if deemed necessary
     3. In the setting of an aortic dissection, access into the true lumen throughout the length of the aorta must be obtainable

Arch Arm Protocol

1. General Inclusion Criteria (Must meet ALL of the following):

   * Life expectancy greater than 2 years
   * Suitable arterial anatomy
   * Absence of systemic disease or allergy that precludes an endovascular repair
   * Capable of giving informed consent and willingness to comply with follow up schedule
   * Patient is considered high or prohibitive risk for open surgical repair of the ascending aneurysm or dissection
2. Anatomic Inclusion Criteria

   * Must meet ALL of the following:

     1. Aneurysm of the ascending aorta or aortic arch/proximal descending thoracic aorta that is >5.5cm or is considered to be at high risk for rupture or dissection given the morphologic characteristics of the aneurysm (or diverticulum).
     2. Proximal aortic fixation zone:

        1. Native aorta or surgical graft (If surgical graft in ascending aorta, the angulation within the graft must be <90 degrees)
        2. Diameter: 20-42mm
        3. Proximal neck length ≥10mm
        4. Ascending aortic length >50mm
        5. Must occur distal to coronary arteries and any coronary artery bypass grafts that are considered patent and necessary for proper cardiac perfusion
     3. Distal aortic fixation zone:

        1. Native aorta or surgical graft
        2. Diameter: 20-42mm
        3. Distal neck length ≥10mm
     4. Supra-aortic trunk (brachiocephalic) vessels

        1. Although the prosthesis will typically have two branches, modifications to the design will allow for a single branch or three branches. Thus, it is generally planned that at least one extra-anatomic bypass graft will be done in conjunction (or in a staged fashion) with the procedure. The two vessels incorporated into the endograft repair would most commonly be the innominate artery and left carotid artery. However, the innominate artery may be coupled with the left subclavian artery in the setting of a bovine arch whereby the flow to the left carotid would come from a left subclavian to carotid bypass. Similarly, the left carotid and subclavian artery may be branched, or simply one vessel branched should specific anatomic limitations exist. In such a situation, multiple extra-anatomic bypasses may be necessary. Thus the inclusion criteria are defined for each artery, yet any combination of arteries may be used for a repair.
        2. Diameter of vessel(s) to be incorporated into endograft

           * Innominate artery: 8-22 mm.
           * Left (or right) common carotid artery: 6-16mm
           * Left (or right) subclavian artery: 5-20mm
           * Length of sealing zone ≥ 10mm
           * Acceptable tortuosity
     5. In the setting of an aortic dissection the following criteria must exist:

        1. Access into the true lumen from the groin and at least one supra-aortic trunk vessel
        2. A sealing zone in the target aorta (or surgical graft) that is proximal to the primary dissection, such that a stent graft would be anticipated to seal off the dissection lumen
        3. A sealing zone in the target supra-aortic trunk vessels that is distal to the dissection, anticipated to seal off the dissection lumen, or surgically created
        4. A true lumen size large enough to deploy the device and still gain access into the target branches
     6. In the setting of a more distal disease, the repair may be coupled with a thoracoabdominal branched device, infrarenal device, and/or internal iliac branch device - typically performed in a staged fashion
     7. Iliac anatomy must allow for the delivery of the arch branch device which is loaded within an 18F-24F sheath. Conduits to the iliac vessels or aorta may be used if deemed necessary.

Thoracoabdominal Arm Protocol

1. General Inclusion Criteria (Must meet ALL of the following):

   * Life expectancy greater than 2 years
   * Suitable arterial anatomy
   * Absence of systemic disease or allergy that precludes an endovascular repair
   * Capable of giving informed consent and willingness to comply with follow up schedule
2. Anatomic Inclusion Criteria

   * Presence of at least one of the following aneurysms is necessary to drive the need for a repair with a fenestrated/branched device:

     1. A thoracoabdominal aortic aneurysm ≥ 5 cm in women and ≥ 5.5 cm in men or suggestive of a high risk of rupture as a result of morphology, growth history or symptoms
     2. A renal artery aneurysm > 20 mm (or twice the diameter of native renal artery)
     3. An SMA aneurysm >30 mm
   * Outside of the "Indications for Use" for commercially available fenestrated or branched endografts approved for use for the treatment of these aneurysms.
   * Proximal neck

     1. Diameter ≤ 40 mm, ≥20 mm
     2. Proximal neck length ≥ 10mm.
     3. The proximal landing zone may be in a prior endograft or a prior surgical graft.
   * Iliac Artery

     1. Diameter ≥ 7 mm (anticipated diameter following balloon angioplasty, stenting, dottoring, or conduit) or ≥ 6 mm for patients receiving an Low-Profile device.
     2. Iliac angulation that will not preclude device delivery or surgical modification of the iliac system
     3. For a bifurcated or aorto-monoiliac prosthesis, iliac implantation sites require ≤ 20 mm in diameter and ≥ 20 mm in length
   * For a straight aorto-aortic prosthesis, distal neck (normal aorta between the aneurysm and iliac bifurcation) ≥ 10 mm in length and ≤ 40 mm in diameter
   * If a hypogastric branch will be used to treat the common iliac aneurysm

     1. The intended common iliac artery is > 20mm in diameter or the aneurysm has morphology concerning for rupture; and
     2. The intended distal fixation site within the internal iliac is ≤ 10mm in diameter.
   * Renal arteries or other visceral vessels arising from the aorta in an orientation that is evident and measurable from cross-sectional imaging (CT or MR)
   * Visceral branch diameters (for incorporated vessels) between 4 mm - 11 mm at the intended distal sealing site (thus distal to a visceral artery aneurysm in such circumstances).
   * Greater than 5 mm of proximal visceral branch length to allow for a seal with the mated device, or the ability to exclude an early branch.
   * In the setting of an aortic dissection the following criteria must exist:

     1. Access into the true lumen from the groin and at least one supra-aortic trunk vessel
     2. A sealing zone in the target aorta (or surgical graft) that is proximal to the primary dissection, such that a stentgraft would be anticipated to seal off the dissection lumen
     3. A sealing zone in the target supra-aortic trunk vessels that is distal to the dissection, anticipated to seal off the dissection lumen, or surgically created
     4. A true lumen size large enough to deploy the device and still gain access into the target branches
   * In the setting of a more proximal disease, the repair may be coupled with an arch-branched device, thoracic aortic endograft, or surgical aortic repair - typically performed in a staged fashion

General Exclusion Criteria

1. Patient can be treated in accordance with the instructions for use with a commercially marketed endovascular prosthesis
2. Pregnancy
3. History of anaphylactic reaction to contrast material with an inability to properly prophylax the patient appropriately
4. Known sensitivity or allergy to materials of construction of the device (including the materials of the LP device).
5. Body habitus that would inhibit X-ray visualization of the aorta
6. Subject had a major surgical or interventional procedure unrelated to the treatment of the aneurysm planned <30 days from the endovascular repair
7. Unstable angina
8. Unwilling to comply with follow up schedule
9. Systemic or local infection that may increase the risk of endovascular graft infection
10. An uncorrectable coagulopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2018-10-25 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | 5 years
  Freedom from death in perioperative and follow up time period
Stroke and TIA | 30 days
  Freedom from peri-operative neurologic event
Aneurysm-related death | 5 years
  Freedom from aneurysm death related to reintervention or incomplete repair

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J Eagleton, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mesnard T, Huang Y, Schanzer A, Timaran CH, Schneider DB, Mendes BC, Eagleton MJ, Farber MA, Parodi FE, Gasper WJ, Beck AW, Sweet MP, Zetterval SL, Lee A, Oderich GS; United States Aortic Research Consortium. Multicenter Prospective Evaluation of Patient Radiation Exposure During Fenestrated-Branched Endovascular Aortic Repair: A Ten-year Experience. Ann Surg. 2025 Feb 18. doi: 10.1097/SLA.0000000000006676. Online ahead of print. PMID 39963789
- [Derived] Oderich GS, Huang Y, Harmsen WS, Tenorio ER, Schanzer A, Timaran CH, Schneider DB, Mendes BC, Eagleton MJ, Farber MA, Gasper WJ, Beck AW, Sweet MP, Lee WA; United States Aortic Research Consortium. Early and Late Aortic-Related Mortality and Rupture After Fenestrated-Branched Endovascular Aortic Repair of Thoracoabdominal Aortic Aneurysms: A Prospective Multicenter Cohort Study. Circulation. 2024 Oct 22;150(17):1343-1353. doi: 10.1161/CIRCULATIONAHA.123.068234. Epub 2024 Jul 11. PMID 38989575
- [Derived] Finnesgard EJ, Beck AW, Eagleton MJ, Farber MA, Gasper WJ, Lee WA, Oderich GS, Schneider DB, Sweet MP, Timaran CH, Simons JP, Schanzer A; United States Aortic Research Consortium. Severity of acute kidney injury is associated with decreased survival after fenestrated and branched endovascular aortic aneurysm repair. J Vasc Surg. 2023 Oct;78(4):892-901. doi: 10.1016/j.jvs.2023.05.034. Epub 2023 Jun 16. PMID 37330702
- [Derived] Aucoin VJ, Motyl CM, Novak Z, Eagleton MJ, Farber MA, Gasper W, Oderich GS, Mendes B, Schanzer A, Tenorio E, Timaran CH, Schneider DB, Sweet MP, Zettervall SL, Beck AW; U.S. Aortic Research Consortium. Predictors and outcomes of spinal cord injury following complex branched/fenestrated endovascular aortic repair in the US Aortic Research Consortium. J Vasc Surg. 2023 Jun;77(6):1578-1587. doi: 10.1016/j.jvs.2023.01.205. Epub 2023 Apr 13. PMID 37059239
- [Derived] Haulon S, Greenberg RK, Spear R, Eagleton M, Abraham C, Lioupis C, Verhoeven E, Ivancev K, Kolbel T, Stanley B, Resch T, Desgranges P, Maurel B, Roeder B, Chuter T, Mastracci T. Global experience with an inner branched arch endograft. J Thorac Cardiovasc Surg. 2014 Oct;148(4):1709-16. doi: 10.1016/j.jtcvs.2014.02.072. Epub 2014 Feb 28. PMID 24685375
- [Derived] Brown CR, Greenberg RK, Wong S, Eagleton M, Mastracci T, Hernandez AV, Rigelsky CM, Moran R. Family history of aortic disease predicts disease patterns and progression and is a significant influence on management strategies for patients and their relatives. J Vasc Surg. 2013 Sep;58(3):573-81. doi: 10.1016/j.jvs.2013.02.239. Epub 2013 Jul 1. PMID 23809203